CLINICAL TRIAL: NCT00714636
Title: Cerebrospinal Fluid Repository
Acronym: CSF
Status: Completed | Type: Observational
Sponsor: Drexel University College of Medicine (Other)
Collaborators: MDA/ALS Center of Hope (Other)
Responsible Party: Sponsor
Organization: Drexel University (Other)
Other Study IDs: Internal-16262
Record Dates: First submitted 2008-07-10; First posted 2008-07-14 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Amyotrophic Lateral Sclerosis; Cerebrospinal Fluid; Neurodegenerative Disease; Motor Neuron Disease
Keywords: Amyotrophic Lateral Sclerosis; Cerebrospinal Fluid; Neurodegenerative Disease; Motor Neuron Disease; Autonomic Nervous System; Neurodegenerative Diseases; Movement Disorders
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Neurodegenerative Diseases; Motor Neuron Disease; Movement Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Cerebrospinal Fluid from Lumbar Puncture.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ALS: Subjects having either definite or probable ALS by El Escorial Criteria.
- Non-ALS: Subjects not having either definite or probable ALS by El Escorial Criteria.

SUMMARY:
The purpose of a CSF repository is to collect samples of spinal fluid from controls and patients with neurologic disorders including but not exclusively ALS, Dementia, CRPS, neuropathies, and other neuromuscular diseases. This CSF repository will allow the use of CSF in biochemical studies of various neurologic diseases. It would also provide a supply of the necessary normal and disease control patients. CSF would be obtained from patients who are undergoing spinal taps for other reasons including diagnosis, treatment, or participation in clinical trials. We are proposing to collect an additional < 3 ml of CSF from a lumbar puncture that is already being performed for diagnostic or therapeutic reasons, in order to store it in our laboratory for use in future research studies. No lumbar punctures will be initiated specifically for this protocol.

DETAILED DESCRIPTION:
The only specific procedures unique to this protocol is the collection of an additional 3ml or less of cerebrospinal fluid from a lumbar puncture already being performed and the collection of clinical information from the patients medical records. Lumbar puncture may be either a research procedure or a standard of care procedure, depending upon the reason for initiating the puncture. We will aliquot the additional fluid into a separate storage container and it will be maintained in the laboratory of Dr. Heiman-Patterson at -70 degrees. Clinical information including age, medical and neurological history, laboratory data, and pathologic information where indicated will be abstracted from the patient chart. All specimens and corresponding clinical information will be labeled with an identification number and sorted by diagnosis. There will be no patient identifying information kept with the specimens. The CSF sample may be used for studies performed by researchers at Drexel University College of Medicine or shared with collaborators. The CSF sample provided will only be used for projects that have approval by the IRB, but subjects will not be notified each time it is used for a study. If CSF sample is still available, consent can be withdrawn at any time by writing a letter to Dr. Heiman-Patterson requesting the withdrawal of the sample.

Researchers will request control and disease specific samples to use in various research studies. There are no DNA studies.

ELIGIBILITY:
Inclusion Criteria:

* Any person undergoing a diagnostic lumbar puncture with a neurologic illness
* Any person undergoing a lumbar puncture as part of anesthesia
* Any person who is undergoing a lumbar puncture for other research purposes such as clinical trials and who has already consented to the lumbar puncture for that purpose.

Exclusion Criteria:

* Anyone who is not undergoing a lumbar puncture for other reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Those undergoing a lumbar puncture for reasons unrelated to this study.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2006-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terry Heiman-Patterson, MD, Principal Investigator — MDA/ALS Center of Hope
Locations (1):
- MDA/ALS Center of Hope, Philadelphia, Pennsylvania, United States